CLINICAL TRIAL: NCT05772221
Title: The Role of Social Determinants in Cardiovascular Health and Vascular Function in a Racial and Ethnic Minority Population at High Risk for Disparities
Brief Title: The Role of Social Determinants in Cardiovascular Health and Vascular Function
Acronym: CVRRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: The University of Texas at Arlington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 022-215
Record Dates: First submitted 2023-03-02; First posted 2023-03-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Social Determinants of Health; Major Depressive Disorder; Cardiovascular Diseases
MeSH Terms: conditions — Depressive Disorder, Major; Cardiovascular Diseases | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interviewer-Administered (Other): Screening assessments to measure social determinants of health in relation to cardiovascular disease.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Screening assessments to measure social determinants of health in relation to cardiovascular disease.

SUMMARY:
This study aims to identify the influence of social determinants of health domains on vascular function in a low income, racial, and ethnic minority population at risk for disparities. We hypothesize that individuals of a lower social economic position and those struggling with depression are at greater risk of cardiovascular disease.

DETAILED DESCRIPTION:
This study aims to identify the influence of social determinants of health domains on vascular function in a low income, racial, and ethnic minority population at risk for disparities. We hypothesize that individuals of a lower social economic position are at greater risk of impairment in the large organ that is responsible for blood movement in the body and artery stiffness. Additional sims include identifying the influence of depression on vascular function and measure the interaction between depression and social determinants of health. We hypothesize that impairment will be greater in individuals with depression than in individuals without. Finally we will compare a comprehensive metabolic project against the social determinants of health and depression, hypothesizing that more severe social determinants of health and depression will increase the risk of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and ability to read.

Exclusion Criteria:

* (1) unable to provide informed consent (e.g., due to acute impairment or psychosis), (2) inability to read, (3) previously enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 1 year
  The PHQ-9 is a self-report measure that assesses the frequency of symptoms on each of the nine DSM-IV criteria for depression for "the last two weeks.". Total scores of 5-9 represent mild depression, 10-14 represent moderate depression, 15-19 represent moderately severe depression, and > 20 represent severe depression.
Generalized Anxiety Disorder-7 (GAD-7) | 1 year
  The GAD-7 is a seven-item self-report scale for identifying the presence of generalized anxiety disorder (GAD) and assessing symptom severity. The items of the GAD- 7 are based on the diagnostic criteria for GAD in the DSM-IV and assess frequency of symptoms over the last two weeks. A score of 10 or greater on the GAD-7 represents a point for identifying cases of GAD. Cut points of 5, 10, and 15 represent mild, moderate, and severe levels of anxiety, respectively.
PTSD Checklist for DSM-V (PCL-5) | 1 year
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Initial research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD across samples.
Perceived Stress Scale | 1 Year
  The Perceived Stress Scale is a 10-item questionnaire widely used to assess stress levels in young people and adults aged 12 and above. It evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable, and overloading over the previous month. Higher scores indicate higher levels of perceived stress.
AAFP Social Needs Screening Tool | 1 year
  This tool is a 15-item questionnaire about a participant's social needs. Social need categories measured by this instrument include housing, food, childcare, employment, education, finances, personal safety, and assistance. Scoring of this instrument highlights areas in an individual's life where there may be a social need.
MacArthur Scale of Subjective Social Status | 1 year
  The MacArthur Scale of Subjective Social Status (MacArthur SSS Scale) is a two-item measure that assesses a person's perceived rank relative to others in their group. Respondents view a drawing of a ladder with 10 rungs, and either read or hear that the ladder represents where people stand in society.
Quality of Life (WHOQOL-BREF) | 1 year
  The WHOQOL-BREF is a 26-item quality of life assessment. It looks at the domains of physical health, psychological, social relationships, and environment. The four domain scores denote an individual's perception of quality of life in each particular domain.
Experiences of Discrimination (EOD) | 1 year
  The EOD is a short self-report instrument. It looks at individuals self-reported experiences of discrimination. Experiences of discrimination categories measures by this instrument include worry questions, global questions, filed complaints, major discrimination, day-to-day unfair treatment, and response to unfair treatment.
WHODAS 2.0 (World Health Organization Disability Assessment Schedule) | 1 year
  The WHODAS is a 36-item version, self- administered assessment. This measure assesses disability across dix domains, including understanding and communicating, getting around, self-care, getting along with people, lie activities, and participation in society.
Social Isolation | 1 year
  Is a 3-item scale used to assess feelings of loneliness or social isolation. Each item has a minimum score of 1 and a maximum score of 3. The higher scores indicate a greater degree of loneliness.
Adverse Childhood Experiences (ACE) | 1 year
  ACE is a 10-item measure used to measure childhood trauma. This questionnaire assesses 10 types of trauma, 5 being personal, physical abuse, verbal abuse, sexual abuse, physical neglect, and emotional neglect and 5 related to family members.
Pittsburgh Sleep Quality Index (PSQI) | 1 year
  PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a one-month period. This measure assesses the following subcategories, sleep quality, latency, duration, habitual sleep efficiency, disturbances use of sleep medication, and daytime dysfunction.
International Physical Activity Questionnaire (IPAQ) | 1 year
  The IPAQ is a 27-item long form, assessing physical activity over the last 7 days. This measure looks at job-related physical activity, transportation physical activity, housework, house maintenance, and caring for family, recreation, sport, and leisure-time physical activity, and time spent sitting.
Connor-Davidson Resilience Scale (CD-RISC-10) | 1 year
  CD-RISC-10 is a 10-item self-report scale measuring resilience. This scale measures resilience and how well an individual is equipped to bounce back after stressful events, tragedy, or trauma. Each item has a minimum score of 0 and a maximum score of 4. Total scores range from 0 to 40. A higher score indicates higher resilience.
Tobacco, Alcohol, Prescription drug, and illicit Substance use Electronic Spanish Platform (TAPS-ESP) | 1 year
  TAPS is a two-stage screening and brief assessment tool that first screens the four broad substance abuse categories (tobacco, alcohol, prescription drug misuse, and illicit substances), then branches to the brief assessment in which the individual is assessed for more specific risks related to an expanded array of substances (tobacco, alcohol, cannabis, cocaine, methamphetamines, prescription stimulants, heroin, prescription opioids, sedatives, and other substances).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sanchez, PhD, Principal Investigator — Baylor Scott and White Research Institute
Locations (1):
- Baylor Scott & White Family Health Center at Juanita J. Craft Recreation Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year